CLINICAL TRIAL: NCT07269275
Title: Prognostic Value of HLA Eplet Mismatches for Long-term Kidney Transplant Outcomes
Brief Title: HLA Eplet Mismatches to Predict Long-term Kidney Transplant Outcomes
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: HLAeplet_kidney survival
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant Failure
Keywords: graft survival; kidney function; prediction; kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Human leukocyte antigen (HLA) matching evaluates the degree of compatibility between donors and organ transplant recipients and assesses broad antigen differences that may influence immune responses post-transplant. A refined HLA matching method based on examining clusters of amino acids on HLA molecules, named eplets, has been recently developed. This method identifies immunogenic discrepancies that may not be apparent through traditional HLA matching. In recent years, assessment of HLA eplet mismatches has emerged as a promising strategy to improve immune risk stratification in kidney transplantation, which is crucial for kidney recipients' management and maximizing allograft longevity. Despite its potential, the prognostic value and clinical relevance of HLA eplet mismatches for predicting long-term kidney allograft failure has not been robustly demonstrated.

In this study, the investigators aim to investigate whether HLA eplet mismatches may represent a relevant clinical tool for patient risk stratification and prediction of long-term allograft failure beyond standard clinical, histological and immunological parameters for monitoring in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased donor kidney recipients transplanted after 2004
* Kidney recipients older than 18 years of age
* Kidney recipients with available HLA genotyping data

Exclusion Criteria:

* Combined transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients from seven European referral centers
Sampling Method: Non-Probability Sample
Enrollment: 5525 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Kidney allograft failure | Up to 10 years after kidney transplantation

SECONDARY OUTCOMES:
Added prognostic value | Up to 10 years after kidney transplantation
  Added prognostic value of HLA eplet mismatches over standard of care monitoring of kidney transplant recipients based on clinical, histological, immunological parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Translational Research Center for Organ Transplantation, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demir Z, Raynaud M, Divard G, Louis K, Truchot A, Niemann M, Ponsirenas R, Aubert O, Del Bello A, Hertig A, Anglicheau D, Dale B, Kamar N, Mangiola M, Zeevi A, Lefaucheur C, Loupy A. Impact of HLA evolutionary divergence and donor-recipient molecular mismatches on antibody-mediated rejection of kidney allografts. Nat Commun. 2025 Jul 1;16(1):5692. doi: 10.1038/s41467-025-60485-y. PMID 40592858
- [Background] Loupy A, Aubert O, Orandi BJ, Naesens M, Bouatou Y, Raynaud M, Divard G, Jackson AM, Viglietti D, Giral M, Kamar N, Thaunat O, Morelon E, Delahousse M, Kuypers D, Hertig A, Rondeau E, Bailly E, Eskandary F, Bohmig G, Gupta G, Glotz D, Legendre C, Montgomery RA, Stegall MD, Empana JP, Jouven X, Segev DL, Lefaucheur C. Prediction system for risk of allograft loss in patients receiving kidney transplants: international derivation and validation study. BMJ. 2019 Sep 17;366:l4923. doi: 10.1136/bmj.l4923. PMID 31530561